CLINICAL TRIAL: NCT01278303
Title: Covered Cheatham Platinum Stents for the Prevention or Treatment of Aortic Wall Injury Associated With Coarctation of the Aorta
Brief Title: Covered CP Stents for the Prevention or Treatment of Aortic Wall Injury Associated With Coarctation of the Aorta
Acronym: COASTII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Harvard University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G060057a; RFD003898A (Other Grant/Funding Number: Food and Drug Administration)
Record Dates: First submitted 2010-08-02; First posted 2011-01-17 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2016-02

CONDITIONS: Aortic Coarctation
Keywords: Coarctation; Aorta
MeSH Terms: conditions — Aortic Coarctation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment of Aortic Wall Injury (Other): Repair of aortic wall injury with covered CP Stents
  Interventions: Device: Treatment of Aortic Wall Injury

INTERVENTIONS:
Device: Treatment of Aortic Wall Injury — A Cheatham covered platinum stent will be implanted in the Descending aorta to repair coarctation of the aorta in qualified patients.

SUMMARY:
Coarctation of the aorta (CoA) is a congenital abnormality producing obstruction to blood flow through the aorta. Coarctation can occur in isolation, in association with bicuspid aortic valve or with major cardiac malformations. CoA accounts for 5-8% of the 8/1000 (4-6/10,000) children born with congenital heart disease. Most CoA is newly diagnosed in childhood; < 25% recognized beyond 10 yrs.

CoA is mostly repaired in childhood by surgery or by balloon catheter dilation. Recurrence rates range from 5-20%. Recurrence is often not recognized until adolescence. Balloon expandable stents have become the predominant therapy in the USA and Europe for CoA treatment in this age group. There are no FDA approved stents for this use. Biliary stents are currently being used off label. Enrollment into a trial of bare metal Cheatham Platinum (CP) Stents, designed for use in CoA, is completed. The Coarctation of the Aorta Stent Trial (COAST) aims to confirm safety and efficacy of CP Stent for native and recurrent CoA.

There are CoA patients with clinical situations that place them at high risk of aortic wall injury during bare metal stenting. Extreme narrowing, genetic aortic wall weakness and advanced age are examples. Patients may present with aortic wall injury (aneurysm) related to prior CoA repair. The occurrence after surgical repair is 3-4% and after balloon dilation 10-20%. Repair of these aneurysms is surgically challenging. The use of fabric-covered CP Stents to prevent or repair aortic wall injury has become the treatment of choice in Europe and recently in the US through the FDA Compassionate Use process. There are no alternative devices available in the US. COAST II will test safety and efficacy of Covered CP Stents to repair or prevent aortic wall injury associated with CoA.

Funding Source-FDA OOPD

DETAILED DESCRIPTION:
There are no prior trials of preventing or treating aortic injury associated with CoA and thus no basis for comparison. A single outcome assessment will not suffice since patients can receive a device for either indication. A 3-category Severity of Illness Scale (SIS) was developed based on clinical judgment of a panel of pediatric cardiologists and reviewed by a Data & Safety Monitoring Board (DSMB) and the FDA Office of Device Evaluation. Five levels of severity have been defined for each of the 3 illness categories, including: Upper extremity hypertension, Upper to lower extremity pressure difference, and Severity of aortic wall injury. The DSMB will assign a level of illness from the SIS for each patient at baseline and one year follow up. Improvement by at least one level will indicate clinical importance. Safety is evaluated by identifying adverse events and comparing their occurrence to surgical repair of CoA in similar age groups reported in the medical literature.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria for use of a Covered CP Stent:

Native or recurrent aortic coarctation* associated with ONE OR MORE of the following:

1. Acute or chronic aortic wall injury, or
2. Nearly atretic descending aorta to 3 mm or less in diameter, or
3. Genetic Syndromes associated with aortic wall weakening. Individuals with genetic syndromes such as Marfan Syndrome, Turner's Syndrome or familial bicuspid aortic valve and ascending aortic aneurysm

   * The significance of aortic obstruction is left to the judgment of the participating investigator.

indications might include mild resting aortic obstruction associated with:

* Exercise related upper extremity hypertension;
* Severe coarctation with multiple and/or large arterial collaterals;
* Single ventricle physiology
* Left ventricular dysfunction
* Ascending aortic aneurysm

  + Aortic wall injury might include:
* Descending aortic aneurysm
* Descending aortic pseudo-aneurysm
* Contained aortic wall rupture
* Non-contained rupture of the aortic wall

Exclusion Criteria:

1. Patient size too small for safe delivery of the device. The absolute lower limit for inclusion under this protocol is 20 kg. However, serious femoral artery injury can occur in small patients, particularly those in the 20-30 kg range and this risk must be reviewed in detail with parents or guardians of children in this weight range.
2. Planned deployment diameter less than 10 mm or greater than 22 mm
3. Location requiring covered stent placement across a carotid artery*
4. Adults lacking capacity to consent
5. Pregnancy

   * crossing or covering of a subclavian artery is acceptable in certain situations, but only after alternative treatments have been considered.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Moore, MD, Principal Investigator — Rady Children's Hospital; John F Rhodes, MD, Principal Investigator — Nicklaus Children's Hospital f/k/a Miami Children's Hospital; Thomas Jones, MD, Principal Investigator — Seattle Children's Hospital; Lisa Bergersen, MD, Principal Investigator — Boston Children's Hospital; Julie A Vincent, MD, Principal Investigator — Morgan Stanley Children's Hospital; Allison Cabalka, MD, Principal Investigator — Mayo Clinic; Henri Justino, MD, Principal Investigator — Baylor College of Medecine, Texas Children's Hospital; Thomas Forbes, MD, Principal Investigator — Children's Hospital of Michigan; Jonathan Rome, MD, Principal Investigator — Children's Hospital of Philadelphia; Joshua Kanter, MD, Principal Investigator — Children's National Research Institute; Phil Moore, MD, Principal Investigator — University of California, San Francisco; Russel Hirsch, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Jacqueline Kreutzer, MD, Principal Investigator — University of Pittsburgh; Thomas Zellers, MD, Principal Investigator — Children's Medical Center Dallas; Lourdes Prieto, MD, Principal Investigator — The Cleveland Clinic; Gregory Fleming, MD, Principal Investigator — Duke University; Dennis Kim, MD, Principal Investigator — Children's Healthcare of Atlanta; John Cheatham, MD, Principal Investigator — Nationwide Children's Hospital; Gregory A Fleming, MD, Principal Investigator — Duke University
Locations (19):
- United States (19):
  - Rady Children's Hospital and Health Center, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Miami Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Children's Hospital of New York - Presbyterian, New York, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - Baylor College of Medicine, Texas Children's Hospital, Houston, Texas
  - Children's Hospital and Regional Medical Center, Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Individual patient data is confidential and not shared.

REFERENCES:
- [Derived] Holzer RJ, Gauvreau K, McEnaney K, Watanabe H, Ringel R. Long-Term Outcomes of the Coarctation of the Aorta Stent Trials. Circ Cardiovasc Interv. 2021 Jun;14(6):e010308. doi: 10.1161/CIRCINTERVENTIONS.120.010308. Epub 2021 May 27. PMID 34039015

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment of Aortic Wall Injury
Started | 82
Completed | 82
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment of Aortic Wall Injury
Number analyzed (Participants) | 82
Age, Continuous [Median (Full Range); unit: years] | 18 [6 to 67]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41
  Between 18 and 65 years | 38
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 52
Region of Enrollment [Number; unit: participants]
  United States | 82

OUTCOME MEASURES:

1. Primary Outcome: Study Participants With Grade 4 or 5 in Degree of Aortic Wall Injury (AWI) and/or Aortic Arch Obstruction Without Clinical Worsening
Description: Severity of Illness Scale (SIS) improvement increase of at least 1 grade from baseline to 12 month follow-up
  SIS is divided into 3 conditions & 5 grades of severity: 1 = worst (reserved for AWI) , 5 = best) C1 Upper Extremity Systolic Blood Pressure (SBP) 2- > 159 mmHg or any hpn on >2 medications 3- 140-159 mmHg or elevated SBP on >2 medications 4- 130-139 mmHg or normal SBP on >2 medications 5- <130 mmHg on 0-2 meds
  C2 Upper Extremity to Lower Extremity SBP difference 2- >59 mmHg 3- 30-59 mmHg 4- 15-29 mmHg 5- <15 mmHg
  C3
  Aortic Wall Injury severity levels:
  1. Uncontained rupture or large aneurysm
  2. Contained rupture or stable large aneurysm
  3. Small contained rupture or moderate aneurysm
  4. Acute, but stable AWI or small aneurysm
  5. No injury or minor aortic wall irregularity not in need of treatment.
     * Grades for conditions represent comparable degrees of illness (0 worst, 5 best) -Grade 0 denotes death related to coarctation or study therapy
Time Frame: Baseline and 12 months
Population: Participants available for analysis at one year
Measure: Number; unit: participants
Arm/Group | Treatment of Aortic Wall Injury
Number analyzed (Participants) | 69
participants | 55

2. Secondary Outcome: Secondary Efficacy Outcomes - 1 Year
Description: Secondary Efficacy Outcomes
  At One Year: (A) Number of participants with arm-leg systolic blood pressure (SBP) differences <15 mmHg and (B) Number of participants with normal or only mildly elevated SBP, no more than mild arm-leg SBP, no clinically significant residual aortic wall injury AND no worsening in any of these three categories
Time Frame: 1 years
Measure: Number; unit: participants
Arm/Group | Treatment of Aortic Wall Injury
Number analyzed (Participants) | 82
participants
  (A) arm-leg SBP difference <15 mmHg | 54
  (B) Good clinical status at 1 yr w/o worsening | 55

3. Secondary Outcome: Secondary Safety Outcomes - Adverse Events
Description: Secondary Safety Outcomes
  The proportion of patients experiencing any serious or somewhat serious adverse event related to the stent or implant procedure by 24 months follow up, such as: new aortic wall injury within the region of covered CP Stent implantation, stent malposition, stent fracture, aortic wall aneurysms (early or late), or restenosis requiring reintervention, arterial access site injury, bleeding, etc.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment of Aortic Wall Injury
Number analyzed (Participants) | 82
percentage of participants
  Serious Adverse Events | 1.2
  Somewhat Serious Adverse Events | 11

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment of Aortic Wall Injury
Serious Adverse Events (participants affected / at risk) | 1/82
Other Adverse Events (participants affected / at risk) | 38/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment of Aortic Wall Injury (N=82)
Aortic Wall Injury (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment of Aortic Wall Injury (N=82)
Arterial Wall Injury (Cardiac disorders) | 2 (2)
Aortic Wall Injury (Cardiac disorders) | 4 (4)
Infection (Infections and infestations) | 1 (1)
Pain or Discomfort (General disorders) | 8 (8)
Neurologic Injury (Nervous system disorders) | 2 (2)
Device Specific (Cardiac disorders) | 8 (8)
Non-Classified (Cardiac disorders) | 2 (2)
Arrhythmia (Cardiac disorders) | 2 (2)
Bruising or Hemorrhage (Blood and lymphatic system disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No